CLINICAL TRIAL: NCT07292831
Title: Geranium Inhalation Aromatherapy: An Alternative Therapy to Alleviate Nausea & Vomiting in Cancer Patients Undergoing Chemotherapy
Brief Title: Geranium Inhalation Aromatherapy for Reducing Nausea and Vomiting in Cancer Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Muhammadiyah Surakarta (Other)
Responsible Party: Principal Investigator, Fahrun Nur Rosyid, Head of Quality Assurance Group, Universitas Muhammadiyah Surakarta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMS-GERANIUM-RCT2025
Record Dates: First submitted 2025-11-23; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting (CINV); Cancer
Keywords: Cancer; Chemotherapy; Geranium Aromatherapy; Nausea; Vomiting
MeSH Terms: conditions — Vomiting; Neoplasms; Nausea | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups: a geranium aromatherapy group and a control group without aromatherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Geranium Aromatherapy (Experimental): Participants in this arm received geranium essential oil inhalation aromatherapy during chemotherapy. The aromatherapy was administered by allowing patients to inhale geranium essential oil through a controlled inhalation method. This intervention was provided during the chemotherapy session, and nausea/vomiting levels were assessed before and 12 hours after chemotherapy using the Index of Nausea, Vomiting, and Retching (INVR).
  Interventions: Other: Geranium Inhalation Aromatherapy
- Control (No Aromatherapy) (No Intervention): Participants in this arm did not receive any aromatherapy or additional supportive intervention. They underwent chemotherapy according to the standard hospital protocol. Nausea and vomiting were assessed at baseline and 12 hours after chemotherapy using the Index of Nausea, Vomiting, and Retching (INVR).

INTERVENTIONS:
Other: Geranium Inhalation Aromatherapy — Participants received inhalation aromatherapy using geranium essential oil (Pelargonium graveolens). The essential oil was administered through controlled inhalation during the chemotherapy session. Patients inhaled the aroma directly, allowing olfactory stimulation intended to reduce nausea and vomiting. The intervention was applied according to a standardized protocol, and nausea/vomiting were assessed before and 12 hours after chemotherapy using the Index of Nausea, Vomiting, and Retching (INVR).
  Other Names: Geranium Essential Oil; Aromatherapy with Geranium Oil
  Arms: Geranium Aromatherapy

SUMMARY:
Chemotherapy-induced nausea and vomiting (CINV) remain among the most distressing side effects experienced by cancer patients and can significantly affect treatment tolerance and quality of life. Geranium essential oil has been proposed as a complementary, non-pharmacological therapy that may help reduce nausea and vomiting through its calming and antiemetic properties.

This randomized controlled trial aims to evaluate the potential effectiveness of geranium inhalation aromatherapy in reducing nausea and vomiting among cancer patients undergoing chemotherapy. Ninety participants undergoing intravenous chemotherapy will be enrolled and randomly assigned to either the geranium aromatherapy group or the control group. The intervention group will receive inhalation of geranium essential oil, while the control group will receive no aromatherapy.Nausea and vomiting will be measured using the validated Index of Nausea, Vomiting, and Retching (INVR) before chemotherapy and 12 hours afterward. This study is designed to explore whether geranium inhalation aromatherapy may serve as a supportive complementary therapy to enhance comfort and overall quality of life for patients undergoing chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy is a primary treatment modality for many types of cancer but is frequently accompanied by adverse effects, particularly nausea and vomiting. These symptoms are triggered by complex interactions between neurotransmitters and receptors in both the gastrointestinal and central nervous systems. Although antiemetic medications have improved over the years, many patients continue to experience discomfort that negatively affects their quality of life. Complementary therapies such as aromatherapy are increasingly explored as supportive approaches to help alleviate these symptoms. Geranium essential oil (Pelargonium graveolens) possesses calming, anti-inflammatory, and potential antiemetic properties. Inhalation aromatherapy is thought to reduce nausea by stimulating olfactory pathways associated with relaxation and autonomic regulation. This study aims to investigate the potential benefit of geranium inhalation aromatherapy as an adjunct to standard chemotherapy care. This randomized controlled trial (RCT) involves 90 cancer patients undergoing intravenous chemotherapy at a public hospital in Surakarta, Indonesia. Participants are selected through simple random sampling. Inclusion criteria include patients aged under 65 years, with a BMI of 18.5-22.9 kg/m², receiving chemotherapy regimen 1, and willing to provide informed consent. Participants will be randomized into two groups: a treatment group receiving geranium inhalation aromatherapy and a control group receiving no aromatherapy. Baseline demographic and clinical characteristics-including age, gender, education level, occupation, body mass index, duration of illness, cancer stage, hemoglobin levels, leukocyte and platelet counts, kidney function, liver function, and chemotherapy status-will be recorded to ensure comparability between groups. Geranium aromatherapy will be administered through inhalation, a method known to deliver rapid olfactory stimulation and promote relaxation. Nausea and vomiting will be assessed using the Index of Nausea, Vomiting, and Retching (INVR), a reliable and widely used instrument for evaluating chemotherapy-related gastrointestinal symptoms. Measurements will be collected at baseline and 12 hours after chemotherapy. This study is expected to provide additional insight into the feasibility, safety, and potential role of aromatherapy-specifically geranium essential oil-in supporting the management of chemotherapy-induced nausea and vomiting as part of a holistic approach to cancer care.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with cancer.
2. Currently undergoing intravenous chemotherapy regimen 1.
3. Aged under 65 years.
4. Body Mass Index (BMI) between 18.5 and 22.9 kg/m².
5. Able and willing to provide informed consent.
6. Able to communicate and follow study instructions.

Exclusion Criteria:

Known allergy or sensitivity to essential oils or fragrances

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Nausea and Vomiting Score (INVR) | Baseline to 12 hours after chemotherapy
  The primary outcome is the change in nausea, vomiting, and retching severity measured using the Index of Nausea, Vomiting, and Retching (INVR). INVR scores are collected before chemotherapy (baseline) and 12 hours after chemotherapy. The measure evaluates the effectiveness of geranium inhalation aromatherapy in reducing chemotherapy-induced nausea and vomiting.

SECONDARY OUTCOMES:
Incidence of Chemotherapy-Induced Nausea and Vomiting (CINV) | 12 hours after chemotherapy
  The secondary outcome is the proportion of participants experiencing nausea and vomiting after chemotherapy, assessed using INVR categorical scores. This measure compares differences in symptom incidence between the geranium aromatherapy group and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Faculty of Health Sciences FIK UMS, Principal Investigator — Universitas Muhammadiyah Surakarta
Locations (1):
- RSUD Dr. Moewardi Surakarta, Surakarta, Centre Java, Indonesia

IPD SHARING:
Plan to Share IPD: No